CLINICAL TRIAL: NCT05662345
Title: ACT-MBC: A Prospective Observational Impact Study of Circulating Tumor Cells (CTCs) in Metastatic Breast Cancer
Brief Title: ACT-MBC: A Study of Circulating Tumor Cells (CTCs) in Metastatic Breast Cancer (MBC)
Acronym: ACT-MBC
Status: Active, not recruiting | Type: Observational
Sponsor: Menarini Silicon Biosystems, INC (Industry)
Collaborators: Medex15 (Industry)
Responsible Party: Sponsor
Other Study IDs: ACT-MBC
Record Dates: First submitted 2022-12-14; First posted 2022-12-22 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cell-Free DNA (cfDNA)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Diagnostic Test: CellSearch Circulating Tumor Cells — Serial CTC enumeration

SUMMARY:
ACT-MBC prospectively assesses the impact of CTCs on treatment decisions, response assessment and prognosis in MBC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Invasive breast cancer with radiographic and/or clinical evidence of advanced metastatic or unresectable disease
2. ER+/HER2- patients prior to starting 2nd line therapy or beyond OR ER/Progesterone Receptor (PR)/HER2-negative (Triple Negative) patients prior to starting any line of therapy
3. Measurable and/or non-measurable disease is allowed
4. Male or female breast cancer is allowed
5. Age > 18 years
6. Willingness to provide mandatory blood specimens
7. Willing to return to enrolling institution for follow up imaging at least once

Exclusion Criteria:

1. Life expectancy of ≤ 6 months
2. Inability to provide blood samples based on the judgment of the treating provider

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Advanced/metastatic breast cancer of following subtypes/lines of systemic therapy in metastatic setting:
  * Estrogen Receptor (ER)+/Human Epidermal growth factor Receptor 2 (HER2) - patients prior to starting 2nd line or later therapy
  * Triple Negative (TN) patients prior to starting any line of systemic therapy
Sampling Method: Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2022-12-12 (Actual); Primary Completion 2025-10-15 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
To prospectively evaluate the impact of CellSearch CTCs on treatment decisions and response assessment in MBC patients | 3 to 4 months
  Assessing proportion of providers that find CellSearch CTCs helpful in determining response to therapy in each unique patient (Questionnaire #2).

SECONDARY OUTCOMES:
Assess barriers and receptiveness of providers in using CTCs in clinical practice | 18 months
  Assessing provider perception of the general usefulness of CTC in pre and post-intervention surveys (Questionnaire #1 and #3)
Evaluate if CTC results correlate with response assessment and disease progression defined by standard of care imaging | 18 months
  Compare baseline and on treatment serial CTCs assessment to identify correlations with first restaging studies and with progression free survival

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Mayo Clinic Health System Albert Lea, Albert Lea, Minnesota
  - Mayo Clinic Health System Mankato, Mankato, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - MCHS Eau Claire, Eau Claire, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided